CLINICAL TRIAL: NCT02306239
Title: the Surgical Intensive Care Unit
Brief Title: The Effect of Terlipressin on Intesitnal Function in Septic Shock Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liu ZiMeng (Other)
Responsible Party: Sponsor-Investigator, Liu ZiMeng, surgical intensive care unit, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012A080204018
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Terlipressin; Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Terlipressin; Norepinephrine

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- norepinephrine (Active Comparator): patients received norepinephrine
  Interventions: Drug: Norepinephrine
- terlipressin (Experimental): patients received terlipressin
  Interventions: Drug: Terlipressin

INTERVENTIONS:
Drug: Terlipressin
  Arms: terlipressin
Drug: Norepinephrine
  Arms: norepinephrine

SUMMARY:
Terlipressin becomes a vasopressin for septic shock. But some studies found it may lead to severe intesitnal complications such as intestinal ischemia. The investigators study was designed to find the effect of terlipressin on intestinal function in septic shock patients.

ELIGIBILITY:
Inclusion Criteria:

* septic shock

Exclusion Criteria:

* shock due to other reasons
* diagnosited intesitinal ischemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
intestinal function assessed by abdominal distension, intestinal bleeding, peritonitis, plasma DAO level, enteral nutrition | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: liu zimeng, master, Principal Investigator — the first affiliated hospital of SUMS
Locations (1):
- the First Affiliated Hospital of Sumyetsan University, Guangzhou, Guangdong, China